CLINICAL TRIAL: NCT02064075
Title: Phase 4 Prospective, Randomized, Blinded Study on the Effect of Different Hydration Strategies on Mortality and Changes in Quality of Life of Patients Suffering From Subarachnoid Haemorrhage
Brief Title: The Mortality and Changes in Quality of Life of Patients Suffering From SAH With Different Hydration Strategies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, assistant lecturer anesthesiologist and intensive care specialist, University of Debrecen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6163-1/2013/EKU; DEOEC RKEB/IKEB:3799-2012 (Other: University of Debrecen,RKEB/IKEB)
Record Dates: First submitted 2014-02-09; First posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid hemorrhage; vasospasm; Lactated Ringer's solution; Hydroxyethyl starch solution
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Ringer's Lactate; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxyethyl starch (Active Comparator): 15 ml/kg Lactated-Ringer's and 15-50 ml/kg hydroxyethyl starch solution was given intravenously every day.
  Interventions: Drug: Hydroxyethyl starch
- Lactated Ringer's solution (Active Comparator): 15-50 ml/kg Lactated-Ringer's solution was given intravenously every day.
  Interventions: Drug: Lactated Ringer's solution

INTERVENTIONS:
Drug: Lactated Ringer's solution — 15-50 ml/kg Lactated-Ringer's solution was given intravenously every day until discharge.
  Arms: Lactated Ringer's solution
Drug: Hydroxyethyl starch — 15 ml/kg Lactated-Ringer's and 15-50 ml/kg hydroxyethyl starch solution was given intravenously every day until discharge.
  Other Names: HES 130/0.4
  Arms: Hydroxyethyl starch

SUMMARY:
Purpose:

- Vasospasm and secondary ischemia following subarachnoidal hemorrhage considerably affect the clinical outcome. The purpose of this study is to determine whether crystalloid (Lactated Ringer's solution) or colloid (hydroxyethyl starch) intravenous infusion is more effective in the treatment of subarachnoid hemorrhage (SAH)

Treatment:

- Patients are randomly divided into two groups. Depending on the blood pressure of the patients the members of the first group receive 15-50 ml/kg Lactated-Ringer's solution daily as part of the treatment, while the others 15 ml/kg Lactated-Ringer's and 15-50 ml/kg hydroxyethyl starch solution daily.

Measurements:

* Neurological status of patients will be determined by the NIH Stoke Scale Score and the Glasgow Coma Scale (GCS) on a daily basis.
* The mid-term survival and quality of life are evaluated with Barthel Index and Glasgow Outcome Scale (GOS) 14 and 30 days following admission to our clinic.

Hypothesis:

-The prevalence of vasospasms, the mortality rate and the medium-term quality of life following subarachnoid hemorrhage is improved if patients are treated with intravenous colloid (hydroxyethyl starch) infusion compared to intravenous crystalloid infusion.

DETAILED DESCRIPTION:
Study protocol:

* Upon arrival Computed Tomography Angiography (CTA), or if necessary, a four-vessel cerebral angiography is carried out in case of each patient. Previous medical history is obtained with particular regard to the onset of the symptoms and the premorbid blood pressure values. Afterwards the Hunt-Hess classification of the patients take place. The neurological condition is recorded with the help of the NIH Stroke Scale on a daily basis. An acute or delayed open surgery or endovascular coiling is carried out by either a neurosurgeon or an interventional neuroradiologist as the definitive treatment of the aneurysm.
* Patients are randomized into two groups, either treated with Lactated Ringer's or hydroxyethyl starch solutions. Patients of the Lactated Ringer's are given 15-50 ml/kg/day Lactated Ringer's infusion from the beginning of their enrollment, while members of the other group receive 15 ml/kg Lactated-Ringer's and 15-50 ml/kg hydroxyethyl starch solution daily. The blood pressure should not exceed the 160 mmHg systolic and 110 mm Hg mean value prior to the definitive treatment. After definitive care the target blood pressure is set to ensure a clinically optimal state, which should not above 150% of the premorbid blood pressure, and should not exceed 200/120 mmHg. In order to achieve and maintain these values additional vasoactive drugs (arterenol, dobutrex) could be administered regardless of the group in a maximum dose of 2.5 micrograms/kg/min arterenol, with an additional dose of 10 ug/kg/min dobutrex if necessary, if the sole intake of intravenous solutions are not sufficient. Blood pressure is measured invasively, continuously after the cannulation of the radial artery.
* Neurological status of patients will be determined by the NIH Stoke Scale Score and the Glasgow Coma Scale (GCS) on a daily basis. The mid-term survival and quality of life are evaluated with Barthel Index and Glasgow Outcome Scale (GOS) 14 and 30 days following admission to our clinic.
* The primary outcome measure of the study is the incidence rate of vasospasm in both groups, while secondary outcome measures included 30-day survival, the neurological status and GOS scores after.

ELIGIBILITY:
Inclusion Criteria:

* patients with subarachnoid hemorrhage
* patients with Hunt-Hess grade I-III.

Exclusion Criteria:

* patients with Hunt-Hess grade IV-V.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The incidence of vasospasm | The presence of vasospasm is assessed daily between Day 1 and Day 14 in average (plus or minus 5 days) after SAH has occured
  The presence of vasospasm is assessed with the help of a transcranial doppler device. Vasospasm is diagnosed if the mean blood flow velocity in the middle cerebral artery is higher than 120 cm/s (centimeter/second)

SECONDARY OUTCOMES:
30-day survival | 30 days after the incidence of SAH
Glasgow Outcome Scale | 30 days after the incidence of SAH
Barthel Index of Activities of Daily Living | 30 days after the incidence of SAH
National Institutes of Health Stroke Scale | 30 days after the incidence of SAH

OTHER OUTCOMES:
Noradrenalin need | 30 days after the incidence of SAH
  The overall noradrenalin need during hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Csilla Molnár, Md, PhD, Principal Investigator — University of Debrecen Medical and Health Science Center Department of Anesthesiology and Intensive Care 4032-Debrecen, Nagyerdei krt 98. Hungary Tel/fax: +36-52-255-347
Locations (1):
- University of Debrecen Medical and Health Science Center Department of Anesthesiology and Intensive Care, Debrecen, Hungary

REFERENCES:
- [Derived] Gal J, Fulesdi B, Varga D, Fodor B, Varga E, Siro P, Bereczki D, Szabo S, Molnar C. Assessment of two prophylactic fluid strategies in aneurysmal subarachnoid hemorrhage: A randomized trial. J Int Med Res. 2020 Jul;48(7):300060520927526. doi: 10.1177/0300060520927526. PMID 32689849